CLINICAL TRIAL: NCT02101931
Title: A Laser Detection for Bladder Cancer by (Photodynamic) Spectra of Urine
Acronym: ALA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Princess Al-Johara Al-Ibrahim Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: E-13-1019; 14/4028/IRB (Registry Identifier: Institutional Review Board)
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Transitional Cell Carcinoma of the Bladder
Keywords: Bladder Cancer; Laser Diagnosis; Amino levulinic Acid; Photodynamic Detection; spectra of urine
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Urine spectral analysis (Experimental): The patient must drink water then the urine will be collected after 4, 8 and 12 hours of taking Amino levulinic Acid and the samples will be analyzed by photodynamic diagnostic procedure. Amino levulinic Acid gets metabolized into certain types of porphyrins which selectively bind on to the tumor tissues (for a longer time than the normal tissues).The above samples is taken in a four side polished quartz cuvette of 1cmx1cmx4cm and put into the table top spectral scan. This consists of a 5 mw, blue diode laser, of 405nm wavelength. The collimated laser beam falls on the urine sample and excites fluorescence and Raman signals from the porphyrin molecules which have been metabolized from the oral administration of Amino levulinic Acid.
  Interventions: Drug: Amino levulinic Acid

INTERVENTIONS:
Drug: Amino levulinic Acid — The bladder cancer patients is required to swallow a chemical called Amino levulinic Acid, about 10mg/kg body weight. 5ml of blood and one urine samples will be taken before using Amino levulinic Acid. The patient must drink water then the urine will be collected after 4, 8 and 12 hours of taking ALA and the samples will be analyzed by photodynamic diagnostic procedure. ALA gets metabolized into certain types of porphyrins which selectively bind on to the tumor tissues (for a longer time than the normal tissues).
  Other Names: Gliolan; Levulan; Levulan Kerastick

SUMMARY:
Research Problem:

Bladder cancer is one of the major health concerns of the world. The present methods of diagnosis are: Ultra sound, Cystoscopy, CT scan and urine cytology. All these are stressful to the patients, particularly Cystoscopy which is commonly employed for the follow up of Bladder cancer patients.

Research Significance:

The present study will employ a new photodynamic diagnostic procedure to quantify a certain cancer specific biomarker called Porphyrin, which selectively binds on to the bladder cancer tissues. In this context the present technique offer viable, very easy and reliable table top instrumentation for diagnosis and continual monitoring of disease regression through urine.

Research Objectives:

* To quantify bladder cancer specific biomarkers such as Porphyrin using photodynamic diagnostic procedure
* To find out whether this technique might be a new and easy tool for bladder cancer diagnosis only by urine.

Research Methodology:

The bladder cancer patients is required to swallow a chemical called ALA (5 Amino levulinic Acid hydrochloride), about 10mg/kg body weight which will play a role of biological indicator. ALA gets metabolized into certain types of porphyrins which selectively bind on to the tumor tissues (for a longer time than the normal tissues). 5ml of blood and one urine samples will be taken before using ALA. The patient must drink water then the urine will be collected after 4, 8 and 12 hours of taking ALA and the samples will be analyzed by photodynamic diagnostic procedure.

DETAILED DESCRIPTION:
Bladder cancer is one of the most common urologic cancers in Saudi Arabia. its cases represent a significant and challenging part in the daily practice for the majority of urologists practicing. The present methods of diagnosis are: Ultra sound, Cystoscopy, CT-scan etc. All these are stressful to the patients, particularly Cystoscopy which is commonly employed for the follow up of Bladder cancer patients.

In recent years, fluorescence cystoscopy, in contrast to conventional white light cystoscopy, has been investigated as a tool to enhance detection of occult papillary lesions and carcinoma in situ. Recent fluorescence photo detection strategies have used 5-aminolevulinic acid (5-ALA); a precursor of heme biosynthesis.

5-Aminolevulinic acid-enhanced cystoscopy does appear to have improved sensitivities in detecting nonmuscle invasive bladder tumors such as carcinoma in situ . Aminolevulinic acid (ALA) may have a role in other applications in surgical oncology based on its ability to discriminate neoplastic tissue from adjacent normal tissue. Aminolevulinic acid is not a photosensitizer, but rather a metabolic precursor of porphyrin, which is a photosensitizer.

The present study will employ photodynamic diagnostic procedure to quantify only in urine a specific cancer biomarker Porphyrin which selectively binds on to the bladder cancer tissues for a longer time than the normal tissues. In this context, the present study will offer viable, very easy and reliable table top instrumentation for diagnosis and continual monitoring of disease regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Urothelial (transitional cell) carcinoma. Early and advanced stages of with transitional cell carcinoma of the bladder before transurethral resection of bladder Tumor (TURBT) .
* Controls: Healthy volunteer's adults matched with age.

Exclusion Criteria:

* Urinary tract infection (UTI) patients
* Cardiac patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Urine spectral profile after four hours | Four hours after taking Amino levulinic Acid
  The bladder cancer patients is required to swallow a chemical called 5 Amino levulinic Acid hydrochloride (ALA), about 10mg/kg body weight. Urine will be collected after four hours of taking Amino levulinic Acid and the samples will be analyzed by photodynamic diagnostic procedure.

SECONDARY OUTCOMES:
Urine spectral profile after eight hours | Eight hours after taking Amino levulinic Acid
  The bladder cancer patients is required to swallow a chemical called 5 Amino levulinic Acid hydrochloride (ALA), about 10mg/kg body weight. Urine will be collected after eight hours of taking Amino levulinic Acid and the samples will be analyzed by photodynamic diagnostic procedure.

OTHER OUTCOMES:
Urine spectral profile after twelve hours | Twelve hours after taking Amino levulinic Acid
  The bladder cancer patients is required to swallow a chemical called 5 Amino levulinic Acid hydrochloride (ALA), about 10mg/kg body weight. Urine will be collected after twelve hours of taking Amino levulinic Acid and the samples will be analyzed by photodynamic diagnostic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Danny M Rabah, Professor, Principal Investigator — College Of Medicine, King Saud University
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in per-reviewed jounal